CLINICAL TRIAL: NCT02970500
Title: Étude Pilote de Phase II Sur l'Effet du méthylphénidate Sur la Fonction Cognitive Des Patientes en rémission d'un Cancer du Sein
Brief Title: Effect of Methylphenidate on Cancer-related Cognitive Impairment
Acronym: CogMet
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We decided to close recruitment in December 2022 as we were having trouble recruiting participants who met our inclusion criteria and the study funding was coming to an end.
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Équipe de Recherche Michel-Sarrazin en Oncologie psychosociale et Soins palliatifs (Unknown); Purdue Pharma LP (Industry); Fondation de l'Hôtel-Dieu de Lévis (Unknown)
Responsible Party: Principal Investigator, Dr Bruno Gagnon, Associate Professor, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-MPH-02-3006
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer Female; Cancer-Related Condition
Keywords: Cognitive impairment; Methylphenidate; Cancer-related cognitive impairment; Mixed method; Phase II study; Breast cancer
MeSH Terms: conditions — Cognitive Dysfunction; Breast Neoplasms | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylphenidate HCl 10Mg SR (Experimental): Participants of the intervention group (n=20) will receive 1 capsule of Methylphenidate HCl 10 mg SR each morning during 14 days during phase 1 and 2 capsules of Methylphenidate HCl 10 mg SR each morning during 14 days during phase 2.
  Interventions: Drug: Methylphenidate HCl 10Mg SR
- Placebo Group (Placebo Comparator): Participants of the control group (n=20) will receive 1 capsule of placebo each morning during 14 days during phase 1 and 2 capsules of placebo each morning during 14 days during phase 2.
  Interventions: Drug: Placebo Group

INTERVENTIONS:
Drug: Methylphenidate HCl 10Mg SR — Methylphenidate HCl 10Mg SR (Phase 1) and Methylphenidate HCl 20Mg SR (Phase 2)
  Arms: Methylphenidate HCl 10Mg SR
Drug: Placebo Group — Placebo
  Arms: Placebo Group

SUMMARY:
Cancer-related cognitive Impairment (CRCI), commonly referred to as "chemo brain" or "brain fog"-impact severely on the Quality of Life (QoL) of cancer survivors. However, it still remains underdiagnosed and challenging to treat. One of the treatment options is the use of psychostimulants such as Methylphenidate (MP), but well-designed clinical trials to test its efficacy are limited. We will conduct a phase II study with a mixed method design to explore the preliminary efficacy of MP to improve cognitive function and QoL in breast cancer patients after treatment with chemotherapy and/or radiotherapy and determine the parameters needed for designing a phase III study.

DETAILED DESCRIPTION:
Objectives: The main objective of this study is to determine the parameters for a phase III study to measure the efficacy of MP in improving CRCI in women with breast cancer who received chemotherapy and/or radiotherapy. In addition, the profile of drug side effects will be estimated. A better understanding of CRCI and its impact on the activities and QoL of the study population is targeted.

Population: The sample will consist of 40 women in remission of non-metastatic breast cancer whose profile meets the following criteria:

1. receiving follow-up at the radio-oncology department of the CHU de Québec-Université Laval or at any other health institutions in Quebec participating in the project;
2. complaining about cognitive impairment;
3. not having any contraindications to the taking of MP or any medical condition that may interfere with his taking and/or any medical condition that could explain the cognitive impairment.

Before study inclusion, the eligibility of these women will be validated by questionnaires and medical records.

Study design: This study will follow the design of a randomized, double-blind, placebo-controlled trial that includes a mixed methodology (convergent design).

Procedures: The study will be divided into two phases. The first phase will start at time T0, before any MP is taken, and will last 14 days (T1). Participants will be assigned to the intervention group, where they will receive 10 mg of MP controlled-release (SR) for 14 days, or the control group where they will receive an identical placebo capsule for 14 days. The second phase begins at T1 and ends 14 days later (T2). This phase will explore a higher dosage. Participants from the intervention group during phase 1 will received an increased dose of MP (20 mg - two capsules) during 14 days whereas participants from the control group will receive two placebo capsules during 14 days.

Measures: Quantitative data. Questionnaires and tests will be used. The effect size calculation will be based on the 'Perceived Cognitive Impairments' (PCI) subscale of the Functional Assessment of Cancer Therapy-Cognitive Function questionnaire (FACT-Cog) test and will be used to determine the required power for a phase III study. Other tests will be explored to assess the sensitivity to measure cognitive changes. Descriptive statistical analysis will be performed. Tests such as the T-Test, χ2 and ANOVA will be used to estimate the degree of improvement of cognitive function by comparing data of the different groups. Qualitative data. Interviews will be conducted with the 40 women included in the study. These interviews will focus on their experience of cognitive deficits before and after taking MP/Placebo at T0 and T2. In order to document the experience of these women and to assess the transferability of the resutls, two methods will be combined to analyze these interviews: an intra-case analysis and an inter-case analysis. Each of the components of the study will answer its main questions independently. However, the data will also be matched (triangulation) to provide a global understanding of the issue and convergence of results when possible.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer stage I, II or III
2. Completed chemotherapy and/or radiotherapy at least 6 months before entering the study
3. Being in remission of breast cancer
4. Complaining of cognitive impairment

Exclusion Criteria:

1. Current or recent use (<2 years) of psychostimulant drugs
2. Women receiving drugs with a potential of interaction with methylphenidate:

   i. Anticoagulants; ii. Antidepressants with the exception of: amitriptyline (≤75mg); citalopram (≤40mg); desipramine (≤75mg); duloxetine (≤60mg); escitalopram (≤20mg); fluoxetine (≤60mg); fluvoxamine (≤150mg); mirtazapine (≤60mg); nortriptyline (≤50mg); trazadone (≤50mg); venlafaxine (≤150mg); vortioxetine (≤20mg); iii. Drugs (cocaine); iv. Erythropoietin; v. Drugs acting on the cerebral dopaminergic system, including drugs that inhibit monoamine oxidase; vi. John's wort, natural medicines for depression or supplements for fatigue.
3. Conditions that may increase the risk of cognitive impairment or toxicity of methylphenidate such as:

   i. Pregnancy and breastfeeding ii. Bipolar status iii. Cerebral tumor or any brain injury iv. Metastatic cancer v. Alcohol addiction vi. Active Major depression vii. Parkinson disease viii. Dementia ix. Epilepsia x. Glaucoma xi. Cardiovascular diseases xii. Auto-immunes and chronic inflammatory disease xiii. Cerebrovascular disease xiv. Narcolepsy xv. Pheochromocytoma xvi. Thyrotoxicosis xvii. Motor tic, Tourette syndrome xviii. Generalized anxiety disorder or panic attacks xix. Living under the same roof as people taking Biphentin® 10 mg capsules (this exclusion criteria is necessary because the placebo capsule is identical to the commercial formulation of Biphentin®) xx. Any other medical criteria, according to the clinical judgment of the principal investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive impairment level | Up to 24 months
  'Perceived Cognitive Impairments' (PCI) subscale of the Functional Assessment of Cancer Therapy-Cognitive Function questionnaire (FACT-Cog) test

SECONDARY OUTCOMES:
Methylphenidate side effects | Up to 24 months
  Tracking and registration of methylphenidate side effects
Methylphenidate effect on fatigue | Up to 24 months
  Fatigue evaluation with a validated questionnaire: Multidimensional Fatigue Inventory (MFI)
Experience of women with cancer-related cognitive impairment in cancer | Up to 24 months
  Semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gagnon, Principal Investigator — Laval University, Centre de recherche du CHU de Québec
Locations (2):
- Canada (2):
  - Hôpital Hôtel-Dieu de Lévis, Lévis, Quebec
  - Centre de recherche du CHU de QUébec, Québec

IPD SHARING:
Plan to Share IPD: No